CLINICAL TRIAL: NCT06416592
Title: Intra-rater and Inter-rater Reliability and Validity of Hand Dynamometer Trunk Flexor, Extensor and Lateral Flexor Muscle Strength Measurements in Patients With Adolescent Idiopathic Scoliosis
Brief Title: Reliability and Validity of Hand Dynamometer Trunk Muscle Strength Measurements in Patients With AIS
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Irem Kurt, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: IUC5
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Scoliosis; Adolescence; Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Rehabilitation; Exercise; Reliability
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intra-rater and inter-rater validity and reliability: Intra-rater and inter-rater validity and reliability of trunk flexion, extension and right-left lateral flexion isometric muscle strength in cases with AIS will be performed with the Lafeyette hand dynamometer device ((Lafayette Manual Muscle Testing System, Lafayette Instrument Co, Lafayette, Indiana). To avoid systematic error, each participant will perform the isometric handheld dynamometer protocol in a random testing order. In order to determine inter-rater reliability, the same hand dynamometer protocol will be applied to each participant by two different assessors on the first day of the test. Participants will be given a 1-hour rest period between evaluators to prevent fatigue in the evaluations to be held on the same day. To determine inter-rater reliability and agreement, participants will be re-evaluated by the same researchers, at the same protocol, place and day, with a 1-week interval to prevent learning effects.

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional complex deformity of the spine characterized by lateral deviation of 10 degrees or more in the frontal plane, rotation in the transverse plane and hypokyphosis in the sagittal plane. It has been reported that in the presence of scoliosis, there is a change in muscle strength of people compared to their healthy peers due to the deterioration of their postural balance. There are many studies in the literature that evaluate the muscle strength of cases diagnosed with scoliosis with objective devices. Among these objective devices, reliability studies on hand dynamometry devices, which are easy to use, portable and cheaper than other devices, have been conducted for different populations. However, no reliability study of the handheld dynamometer device in patients with AIS has been found in the literature. Therefore, the aim of our study is to study the intra-rater and inter-rater reliability and validity of the trunk flexion, extension and lateral flexion muscle strengths of the hand dynamometer device in cases with AIS, which are known to have changes in muscle strength compared to their peers as a result of the change in spinal alignment. After obtaining the demographic information of the cases that meet the inclusion criteria within the scope of the study, the isometric muscle strength of the trunk flexor, extensor and right-left lateral flexor muscles will be evaluated by two different evaluators using a Lafayette hand dynamometer. To avoid systematic error, each participant will perform the isometric handheld dynamometer protocol in a random testing order. In order to determine interobserver reliability, on the first day of the test, the same hand dynamometer protocol will be applied to each participant by two different evaluators, after a 1-hour rest to prevent fatigue. To determine intraobserver reliability and compliance, participants will be re-evaluated by the same researchers at the same protocol, place and day period, 1 week apart to prevent learning effects. This study will reveal the intraobserver and interobserver reliability and validity of the handheld dynamometer device, which can be used in the evaluation of trunk muscle strength for clinicians working with AIS.

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a three-dimensional complex deformity of the spine characterized by lateral deviation of 10 degrees or more in the frontal plane, rotation in the transverse plane and hypokyphosis in the sagittal plane, and is an important public health problem with a global prevalence of 0.47-5.2%. Muscle strength is an important factor in maintaining postural balance in AIS, and it is observed that both clinicians and researchers evaluate the muscle strength of cases with AIS using different objective devices. Objective muscle strength assessment methods include electromyography, hand dynamometry and isokinetic dynamometry. Electromyography devices and isokinetic dynamometers are expensive and their use in the clinic is limited because they are not easily portable. Therefore, it has been shown to be a valid and reliable method to evaluate trunk muscle strength in different populations and pathologies such as healthy adults, healthy athletic individuals, chronic low back pain or hemiplegic patients; The handheld dynamometer device, which has the advantage of being cheaper and more portable than other devices, appears as a suitable option for clinicians to evaluate trunk isometric muscle strength. No reliability studies of hand dynamometer devices have been found in the AIS population. Therefore, our aim in the study is to study the intra-observer and inter-observer reliability and validity of the trunk flexion, extension and lateral flexion muscle strengths of the hand dynamometer device in patients with AIS, who are known to have changes in muscle strength compared to their peers as a result of the change in spinal alignment. This study will reveal the validity of the hand dynamometer device that can be used in the evaluation of trunk muscle strength for clinicians working with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 10-18
* Having been diagnosed with Adolescent Idiopathic Scoliosis by an orthopedic specialist
* Ability to understand instructions
* Volunteering to participate in the study

Exclusion Criteria:

* History of traumatic trunk or pelvic injury
* History of acute, subacute or chronic low back pain or neurological disease
* Having had spinal surgery
* Participating in heavy physical activity at least one day before the test days
* Having experienced any acute situation that could affect muscle strength between the two tests (within 7 days)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent idiopathic scoliosis patients
Sampling Method: Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Isometric trunk flexor strength | Baseline (All rater), after 1 hour (Rater 1) and 1 week (Rater 1)
  Isometric trunk flexor strength, two different test positions were adapted based on current literature. The first position will be measured on the back at 0 degrees of extension, with the knees straight. The dynamometer will be placed below the suprasternal notch of the sternum. Participants will be instructed to place their hand on the opposite acromion. To prevent pelvic rotation, participants will be fixed with the help of a belt from the anterior superior iliac spine and 10 cm above the lateral malleolus. The second position will be measured on the back in a 30 degree flexion position with the knees straight. The dynamometer will be placed below the suprasternal notch of the sternum. Participants will be instructed to place their hand on the opposite acromion. To prevent pelvic rotation, participants will be fixed with the help of a belt from the anterior superior iliac spine and 10 cm above the lateral malleolus.
Isometric trunk extension strength | Baseline (All rater), after 1 hour (Rater 1) and 1 week (Rater 1)
  Isometric trunk extension strength, two different test positions were adapted based on current literature. The first position will be measured face down in 0 degree extension position. The dynamometer will be placed at the height T4. Participants will be instructed to place their hands on their foreheads. Participants will be fixed with the help of a belt from the posterior superior iliac spine and 10 cm above the lateral malleolus to prevent pelvic rotation. The second position will be measured face down in a 30 degree flexion position. The dynamometer will be placed at the height T4. Participants will be instructed to place their hands on their foreheads. Participants will be fixed with the help of a belt from the posterior superior iliac spine and 10 cm above the lateral malleolus to prevent pelvic rotation.
Isometric trunk lateral flexion strength | Baseline (All rater), after 1 hour (Rater 1) and 1 week (Rater 1)
  Isometric trunk lateral flexion strength will be measured in the sitting position. Participants will sit on a chair with their feet not touching the ground and their hips in 90° flexion, and the participant will be fixed with the help of a strap. The dynamometer will be placed at shoulder level. Participants will be instructed to place their hand on the opposite acromion. Trials in which excessive motion (a detectable amount of movement or rotation in the transverse plane) occurs will be rejected and measured as.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Kurt Ulusoy, Principal Investigator — Istanbul University - Cerrahpasa; Elcin Akyurek, Principal Investigator — Istanbul University - Cerrahpasa; İpek Yeldan, Principal Investigator — Istanbul University - Cerrahpasa; Ayse Zengin Alpozgen, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İrem Kurt, Istanbul, Turkey (Türkiye)